CLINICAL TRIAL: NCT05407818
Title: A Phase 1, Open-label, Single Dose Study to Investigate Pharmacokinetics, Safety and Tolerability of JNJ-63733657 in Healthy Chinese Participants
Brief Title: A Study of JNJ-63733657 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR109144; 63733657ALZ1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JNJ-63733657 (Experimental): Participants will receive a single dose of JNJ-63733657 as an intravenous (IV) infusion on Day 1.
  Interventions: Drug: JNJ-63733657

INTERVENTIONS:
Drug: JNJ-63733657 — JNJ-63733657 will be administered as an IV infusion.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of JNJ-63733657 following single intravenous (IV) dose administration in healthy Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy for their age group on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiograms (ECGs) performed at screening. If there are any abnormalities, they must be considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy for their age group on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel including liver enzymes, other specific tests, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI) between 18 and 35 kilograms per meter square (kg/m^2) (inclusive), and body weight greater than 50 kilograms (kg) but less than 80 kg (in order not to exceed the total dose of 5 grams [g] JNJ-63733657) at screening
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 150 millimeters of mercury (mm Hg) systolic, inclusive, and no higher than 90 mm Hg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted. The participant will be considered eligible if any one of the blood pressure assessments within the range of 90-150 systolic and less than 90 diastolic
* Willing and able to adhere to the prohibitions and restrictions specified in the protocol

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Known allergies, hypersensitivity, or suspected intolerance to any biologic medication or known allergies, or clinically significant reactions to human proteins, monoclonal antibodies or antibody fragments, JNJ-63733657 or its excipients
* Taken any disallowed therapies, concomitant therapy before the planned administration of study intervention. The use of medication that is considered not to have any impact on the study results may be allowed after agreement between the investigator and the sponsor's medical monitor
* Received an investigational drug (including vaccines) or used an experimental medical device within 3 months or within a period less than 5 times the drug's half-life, if known, whichever is longer, before the administration of study intervention
* Preplanned surgery or procedures that would interfere with the conduct of the study

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Serum Concentrations of JNJ-63733657 | Up to Week 13
  Serum samples will be analyzed to determine concentrations of JNJ-63733657 using a validated, specific, and sensitive Immunoassay method.

SECONDARY OUTCOMES:
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) by Severity | Up to Week 13
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment. An assessment of severity grade will be made using the following general categorical descriptors: Mild, Moderate, and Severe.
Percentage of Participants with Discontinuations due to AEs | Up to Week 17
  Percentage of participants with discontinuations due to AEs will be reported.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 17
  An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Percentage of Participants with Clinically Significant Changes in Vital Signs | Up to Week 17
  Percentage of participants with clinically significant changes in vital signs (including temperature [axillary], pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Percentage of Participants with Clinically Significant Changes in Electrocardiograms (ECGs) | Up to Week 17
  Percentage of participants with clinically significant changes in ECGs will be reported.
Percentage of Participants with Clinically Significant Changes in Clinical Safety Laboratory Parameters | Up to Week 17
  Percentage of participants with clinically significant changes in clinical safety laboratory parameters (including hematology, chemistry, and urinalyses) will be reported.
Percentage of Participants with Anti-drug Antibodies to JNJ-63733657 | Up to Week 13
  Percentage of participants with anti-drug antibodies to JNJ-63733657 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency